CLINICAL TRIAL: NCT01103401
Title: Ketorolac Plus Tobramycin/Dexamethasone vs. Tobramycin/Dexamethasone After Uneventful Phacoemulsification Surgery
Brief Title: Ketorolac Plus Tobramycin/Dexamethasone Versus Tobramycin/Dexamethasone After Uneventful Phacoemulsification Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veroia General Hospital (Other)
Responsible Party: Department of Ophthalmology, Veroia General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGH-EYE02
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Tobramycin; Tobramycin, Dexamethasone Drug Combination; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobramycin/Dexamethasone (Active Comparator)
  Interventions: Drug: Drug: Tobramycin 0.3% - Dexamethasone 0.1%; Drug: Drug: Tobramycin-Dexamethasone plus Ketorolac tromethamine
- Tobramycin/Dexamethasone plus Ketorolac tromethamine (Active Comparator)
  Interventions: Drug: Drug: Tobramycin 0.3% - Dexamethasone 0.1%; Drug: Drug: Tobramycin-Dexamethasone plus Ketorolac tromethamine

INTERVENTIONS:
Drug: Drug: Tobramycin 0.3% - Dexamethasone 0.1% — one drop four times per day
  Other Names: Tobradex
Drug: Drug: Tobramycin-Dexamethasone plus Ketorolac tromethamine — Tobramycin-Dexamethasone one drop four times per day and Ketorolac tromethamine one drop three times per day
  Other Names: Acular

SUMMARY:
This randomized controlled trial compares two regimens of topical therapy:

* tobramycin 0.3% - dexamethasone 0.1% (TobraDex®, Alcon), one drop four times/day
* combination of tobramycin 0.3% - dexamethasone 0.1% (TobraDex®, Alcon), one drop four times/day, plus Ketorolac tromethamine 0.5% (Acular®, Allergan), one drop three times/day.

Patients are independently assessed by two ophthalmologists. On days 7,14,21,28 patients are evaluated for

* corneal edema
* conjunctival hyperemia
* anterior chamber (Tyndall) reaction.

The investigators purpose was to evaluate the benefit of adding a non-steroid agent to an antibiotic/steroid combination after uneventful phacoemulsification. Adopting a weekly follow-up, to gain insight into the optimal duration of postoperative treatment and to examine whether risk factors for inflammation exist.

DETAILED DESCRIPTION:
Patients were randomized to: i) tobramycin 0.3% - dexamethasone 0.1% one drop qid (TD group, n=72, 28 days) and ii) combination of tobramycin 0.3% - dexamethasone 0.1%, one drop qid, plus Ketorolac tromethamine 0.5%, one drop tid (TD-K group, n=73, 28 days). Patients undergoing vitrectomy due to posterior capsule rupture were excluded. On days 7, 14, 21, 28, the frequency of inflammation-related signs [corneal edema, conjunctival hyperemia, anterior chamber (Tyndall) reaction], as well as the best corrected visual acuity (BCVA) were measured. On day 21, logistic regression was performed to evaluate risk factors for inflammation.

ELIGIBILITY:
Inclusion Criteria:

* phacoemulsification (due to cataract)
* uneventful phacoemulsification surgery

Exclusion Criteria:

* history of intraocular surgery in the operated eye,
* any previous episode of uveitis in the operated eye,
* severe systemic disease (heart failure NYHA stage III of IV, end-stage renal failure, pulmonary failure, patients receiving chemotherapy),
* regular, systemic use of steroid or non-steroid anti-inflammatory drugs during the last three months
* disruption of the anterior lens capsule

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity, corneal edema, Tyndall reaction, redness | 1,7,14,28 post-operative day, Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas E Papazisis, Director, Study Director — leopapazisis@yahoo.gr